CLINICAL TRIAL: NCT02320890
Title: A Study for the Short- and Long-term Improvement of Cognitive Function (Evaluated by PET-CT and SNSB) After Transcranial Direct Current Stimulation in Mild Cognitive Impairment
Brief Title: Study of tDCS for Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Collaborators: Ybrain Inc. (Industry)
Responsible Party: Principal Investigator, Yong An Chung, Professor of Radiology, Catholic University of Korea, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OC14OISI0045
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Mild Cognitive Impairment
Keywords: transcranial direct current stimulation; tDCS; Mild Cognitive Impairment; MCI
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- YBand (YDT-201N) (Experimental): transcranial Direct Current Stimulation (tDCS) application 3 days a week for 12 weeks (total of 36 applications)
  Interventions: Device: YBand (YDT-201N)
- sham-Yband (YDT-201N) (Sham Comparator): sham-tDCS application 3 days a week for 12 weeks (total of 36 applications)
  Interventions: Device: sham-YBand (YDT-201N)

INTERVENTIONS:
Device: YBand (YDT-201N) — transcranial Direct Current Stimulation (tDCS) 2mA for 30 min; 20 sec of ramp-up and -down; left(anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)
  Arms: YBand (YDT-201N)
Device: sham-YBand (YDT-201N) — transcranial Direct Current Stimulation (tDCS) 2mA for 20 sec; left (anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)
  Arms: sham-Yband (YDT-201N)

SUMMARY:
The primary objective of this study is to investigate whether the transcranial direct current stimulation (tDCS) improves the cognitive function in patients with Mild Cognitive Impairment (MCI)

DETAILED DESCRIPTION:
Twenty-four patients were recruited and randomized to receive either real- or sham-tDCS over the left (anode) and right (cathode) dorsolateral prefrontal cortex (DLPFC). Their legally responsible caregivers were provided with mobile tDCS device, and were instructed to use it on the patients at the hospital. 30-minute session of the stimulation were applied 3 times a week for 12 weeks. The patients were evaluated at baseline and at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a subjective memory impairment
* Subjects who have Korean version of Mini Mental Status Examination score 22 or more
* Subjects who have SVLT and RCFT delayed recall test scores lower than 1.5SD
* Subjects who have had other cognitive impairments besides memory
* Subjects who have Seoul-Instrumental Activities of Daily Living score (S-IADL) of 8 or lower
* Subjects who are not dementia of Alzheimer's type
* Subjects who are right-handed
* Subjects who are able to read and write
* Subject or legally responsible caregiver has provided informed consent

Exclusion Criteria:

* Subjects who have a history of stroke and seizures
* Subjects who have any illnesses that may disturb the patients completing the trials, including stroke, Parkinson's disease, type 1 diabetes, uncontrollable high blood pressure, Huntington's disease, cerebral palsy, liver failure, nephritis, encephalitis, meningitis, scleroma, seizures and a treatment ischemic attack.
* Subjects who have neurologic problems on physical examination that cuase memory disturbances
* Subjects who have a history of DSM-IV Axis I disorders
* Subjects who have extremely sensitive skin
* Subjects who have suffered from the cancer in 3 years
* Subjects who have had a cerebrovascular neurosurgery in medical history
* Subjects who have dyspnea in sitting position
* Subjects who have problems with memory, language and problem-solving for 2 hours after the heart attack.
* Subjects who have a history of drug or alcohol abuse (in the past 5 years)
* Subjects who have a history of mental or emotional disorders (in the past 5 years)
* Subjects who have been lapsed into unconsciousness for an hour because of other reasons than general anesthesia
* Subjects who have a history of hospitalization due to head injury
* Subjects who are unable to read even with glasses
* Subject who are unable to understand the conversation due to the hearing defect (even with the hearing aid)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in PET-CT images | from baseline to Week 12

SECONDARY OUTCOMES:
Change in Cognitive function | from baseline to Week 12
  Measured by SNSB
Change in Cognitive function | from baseline to Week 12
  Measured by Korean version of Mini Mental Status Examination (K-MMSE) and Clinical Dementia Rating (CDR)
Change in activities of daily living | from baseline to Week 12
  Measured by B-ADL
Change in Geriatric Depression Scale | from baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Yong-An Chung, M.D., Ph.D., Principal Investigator — Professor, Department of Radiology
Locations (1):
- Incheon St.Mary's Hospital, Incheon, South Korea